CLINICAL TRIAL: NCT05314998
Title: An Open Labelled Phase III Adjuvant Trial of Disease-free Survival in Patients With Resected Pancreatic Ductal Adenocarcinoma Randomized to Allocation of Oxaliplatin- or Gemcitabine-based Chemotherapy by Standard Clinical Criteria or by a Transcriptomic Treatment Specific Stratification Signature
Brief Title: Adjuvant Trial in Patients With Resected PDAC Randomized to Allocation of Oxaliplatin- or Gemcitabine-based Chemotherapy by Standard Clinical Criteria or by a Transcriptomic Treatment Specific Stratification Signature
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: John Neoptolemos (Other)
Collaborators: Molecular Health GmbH (Industry); German Cancer Research Center (Other); Nationales Centrum für Tumorerkrankungen (Unknown); Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other); Institut für Medizinische Biometrie (Unknown)
Responsible Party: Sponsor-Investigator, John Neoptolemos, Prof. Dr. med., Heidelberg University
Organization: Heidelberg University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESPAC-6; AIO-PAK-0121/ass (Other: AIO); 2020-004906-79 (EudraCT Number)
Record Dates: First submitted 2022-03-29; First posted 2022-04-07 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic Ductal Adenocarcinoma; PDAC
MeSH Terms: interventions — Oxaliplatin; Irinotecan; Leucovorin; Fluorouracil; Gemcitabine; Capecitabine

STUDY DESIGN:
Intervention Model Description: Therapeutic intervention of standard adjuvant chemotherapy comprising oxaliplatin- or gemcitabine-based regimens based on standard clinical criteria, compared to selection using a treatment specific signature and prediction model.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Arm A: mFOLFIRINOX or Gem/Cap according to transcriptomic treatment specific signature (Experimental): mFOLFIRINOX-therapy (5-FU, Folinic Acid, Irinotecan, Oxaliplatin) according to individual transcriptomic treatment specific signature or Gem/Cap-therapy (Gemcitabine and Capecitabine) according to individual transcriptomic treatment specific signature
  Interventions: Drug: Oxaliplatin; Drug: Irinotecan; Drug: Folinic acid; Drug: 5-fluorouracil; Drug: Gemcitabine; Drug: Capecitabine
- Control Arm B: mFOLFIRINOX or Gem/Cap according to standard clinical criteria (Active Comparator): mFOLFIRINOX-therapy (5-FU, Folinic Acid, Irinotecan, Oxaliplatin) according to standard clinical criteria or Gem/Cap-therapy (Gemcitabine and Capecitabine) according to standard clinical criteria
  Interventions: Drug: Oxaliplatin; Drug: Irinotecan; Drug: Folinic acid; Drug: 5-fluorouracil; Drug: Gemcitabine; Drug: Capecitabine

INTERVENTIONS:
Drug: Oxaliplatin — 85 mg/m2 D1 over 2 hours every; 14 days, 12 cycles, 24 weeks
Drug: Irinotecan — 150 mg/m2 D1 over 90 minutes to begin 30 min after the Folinic acid infusion is started; every 14 days, 12 cycles, 24 weeks
Drug: Folinic acid — 400 mg/m2 (racemic mixture) (or 200 mg/m2 if L-folinic acid is used), IV infusion over 2 hours; every 14 days, 12 cycles, 24 weeks
Drug: 5-fluorouracil — 2.4 g/m2 IV continuous infusion over 46 hours (1200 mg/m2/ day); every 14 days, 12 cycles, 24 weeks
Drug: Gemcitabine — 1000mg/m2 is given as an IV infusion over 30 minutes; on day 1, 8 and 15 out of 28 days (= 1 cycle); Repeated 6 times (i.e., 6 cycles) for 24 weeks
Drug: Capecitabine — 1660mg/m2/day in two divided doses administered orally for 21 days followed by 7 days' rest (one cycle) for six cycles i.e. 24 weeks

SUMMARY:
This is a multicentre open labelled phase III adjuvant trial of disease-free survival in patients with resected pancreatic ductal adenocarcinoma randomized to allocation of oxaliplatin- or gemcitabine-based chemotherapy by standard clinical criteria (control arm) or by a transcriptomic treatment specific stratification signature or TSS (test arm).

DETAILED DESCRIPTION:
The main purpose and primary objective of the study is to determine whether disease free survival in patients with resected pancreatic ductal adenocarcinoma (PDAC) treated with standard adjuvant chemotherapy regimens (oxaliplatin- or gemcitabine-based), is superior using allocation based on a treatment specific signature (TSS), compared to the same chemotherapy regimens allocated according to standard clinical criteria.

Secondary objectives of the study are to assess overall survival (median, 3 year survival rate), metastasis free survival; survival based on targeted signatures (TSS) in test versus control arms, and survival using targeted therapies initially on relapse compared to standard first-line therapies on relapse.

In addition, ESPAC-6 optional translational research programme will obtain tumor specimens and blodd samples to identify biomarkers that may predict response to chemotherapy or relapse.

ESPAC-6 will also generate a biobank of matched patient-derived organoids (PDOs) to provide an experimentally tractable model system for the development and testing of biomarker-driven personalised therapies.

ESPAC-6 translational research programme, will also develop a longitudinal blood biobank to analyse clinically relevant circulating biomarkers, such as blood proteins, metabolites and/or circulating-free tumour DNA.

ELIGIBILITY:
Inclusion Criteria

1. Histologically proven pancreatic ductal adenocarcinoma including variants, and pancreatic acinar cell carcinoma.
2. Patient had provided tumour tissue at resection for RNAseq.
3. Macroscopically complete resection (R0 or R1 resection).
4. Female and male Patients aged from 18 to 79 years.
5. WHO performance status 0-1.
6. No prior radiotherapy and no previous chemotherapy for pancreatic cancer.
7. Full recovery from surgery and patient able to receive chemotherapy: adequate oral nutrition of ≥ 1500 calories per day and free of significant nausea and vomiting.
8. Adequate hematologic function: Absolute neutrophil count ≥ 1,500 cells/mm3, platelets ≥ 100,000 cells/mm3 and haemoglobin ≥ 8 g/L (transfusion permitted).
9. Serum total bilirubin ≤ 1.5 times the institutional upper limit of normal.
10. Creatinine clearance ≥ 50 mL/min.
11. Patient of child-bearing potential (for female patient: study entry after a menstrual period and a negative pregnancy test) must agree to use highly effective methods of contraception during the study and for 6 months after the last study treatment for women and 6 months for men.
12. Intended interval since surgery between 21 and 84 days at date of randomization.
13. Public or private health insurance cover.
14. Ability of subject to understand character and individual consequences of the clinical trial.
15. Not legally incapacitated.
16. Written informed consent.

Exclusion Criteria

1. Solid pseudopapillary neoplasm, neuroendocrine neoplasm, pancreatoblastoma, bile duct cancer, and ampullary cancer.
2. Distant metastases, including ascites or malignant pleural effusion.
3. Macroscopic incomplete tumour removal (R2 resection).
4. Post-operative CA 19-9 > 180 U / ml before randomization on study.
5. Cardiomyopathy or congestive heart failure, NYHA III-IV or coronary heart disease symptoms.
6. Major comorbidity that may preclude the delivery of treatment or known active infection (HIV or untreated chronic hepatitis B or active hepatitis C) or uncontrolled diabetes.
7. Pre-existing neuropathy, Gilbert's disease or known genotype UGT1A1*28 /*28.
8. Inflammatory disease of the colon or rectum, or intestinal obstruction, or severe postoperative uncontrolled diarrhoea.
9. Known severe dihydropyrimidine dehydrogenase (DPD) deficiency (activity score <1). There are clear guidelines for dose reductions for patients with a score of 1 and 1,5 (2 is normal activity)
10. Pregnancy and lactation.
11. Participation in other clinical trials or observation period of competing trials, respectively.
12. History of hypersensitivity or other known contraindication to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product.
13. Past or current history of other malignancies not curatively treated and without evidence of disease for more than 5 years, except for curatively treated basal cell carcinoma of the skin and in situ carcinoma of the cervix or bladder, or low/intermediate risk prostate cancer (Gleason score ≤7) with normal PSA levels.
14. Any other concurrent antineoplastic treatment including irradiation

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2031-01-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 76 months
  Disease free survival will be defined as time from ramdomisation to disease recurrence (growth or metastasis) or death from any cause all patients fulfilling the in- and exclusion criteria.

SECONDARY OUTCOMES:
Overall survival | 76 months
  Overall survival is defined as the time from randomization to death due to any cause. If a patient is lost to follow up, overall survival time is censored at the time of last contact.
Metastasis free survival | 76 months
  Metastasis free survival is defined as the time from randomization to detection of metastasis or death from any cause. The time of metastasis is defined as the date of metastasis determined and recorded by the Pancreas Tumour Board (Multidisciplinary Team).
  If the patient is eligible for first line therapy the recurrence must be performed by a positive biopsy or cytology.
  If a patient is lost to follow up, metastasis free survival time is censored at the time of last contact.
Overall survival from recurrence | 76 months
  Overall survival is defined as the time from recurrence to death due to any cause. If a patient is lost to follow up, overall survival time is censored at the time of last contact.
Quality of life (QoL EORTC QLQ-C-30) | 76 months
  QoL will be assessed by the EORTC QLQ-C30 questionnaire in its most current version every three months starting from V1.
Safety: (serious) adverse events and Grade 3 and 4 toxicities according to NCI-CTC v.5.0. | 47 months
  Safety assessments will include adverse events. The proportion of grade 3 and 4 toxicity will be compared across treatments using time to event methods and frequency counts. Adverse and serious adverse events are collected throughout the study and will be tabulated and compared between study arms.
  The analysis of all safety endpoints is conducted on the safety set, which contains all patients who received at least one cycle of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: John Neoptolemos, Prof. Dr., Study Director — Universität Heidelberg
Locations (33):
- Germany (28):
  - Universitätsklinikum Aachen, Studienzentrum Viszeralmedizin Klinik für Allgemeine-, Viszeral und Transplatationschirurgie, Aachen
  - Universitätsklinikum Augsburg, III. medizinische Klinik, Augsburg
  - St. Josef-Hospital, Klinikum der Ruhr-Universität Bochum, Abteilung für Hämatologie, Onkologie und Palliativmedizin, Studienambulanz, Bochum
  - Universitätsklinikum Bonn, Chirurgische Abteilung, Bonn
  - DIK Deggendorf, Onkologische Ambulanz, Deggendorf
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Klinik und Poliklinik für Viszeral-, Thorax- und Gefäßchirurgie, Dresden
  - Universitätsklinikum Erlangen, Chirurgische Klinik Zentrum für klinische Studien, Erlangen
  - Universitätsklinikum Frankfurt, Klinik für Allgemein-, Viszeral- und Transplantationschirurgie,, Frankfurt
  - Universitätsklinikum Freiburg, Klinik für Allgemein und Viszeralchirurgie, Abteilung Chirurgie, Freiburg im Breisgau
  - Universitätsklinikum Halle (Saale), Klinik und Poliklinik für Innere Medizin I, Halle
  - Universitätsklinikum Hamburg Eppendort, Zentrum für operative Medizin, Klinik und Poliklinik für Allgemein-, Viszeral- und Thoraxchirurgie, Hamburg
  - Medizinische Hochschule Hannover, Klinik für Gastroenterologie, Hepatologie und Endokrinologie, Hanover
  - Universitätsklinikum Heidelberg, Abteilung für Allgemein-, Viszeral- und Transplantationschirurgie und Nationales Zentrum für Tumorerkrankungen, Medizinische Onkologie, Heidelberg
  - Universitätsklinikum des Saarlandes, Klinik für Innere Medizin II und Klinik für Allgemeine Viszeral Gefäß und Kinderchirurgie, Homburg/Saar
  - Univeristätsklinikum Jena, Jena
  - UKSH Campus Kiel, Medizinische Klinik II, Kiel
  - Universität Leipzig, Medizinische Fakultät, Klinik für Gastroenterologie, Hepatologie, Infektiologie und Pneumologie, Leipzig
  - Universitätsklinikum Schleswig-Holstein, Klinik für Chirurgie, Onkologisches Zentrum Campus Lübeck, Lübeck
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, I. medizinische Klinik, Klinik für Allgemein-, Viszeral- und Transplantationschirurgie, Mainz
  - Universitätsklinikum Mannheim, II. medizinische Klinik, Klinik für Gastroenterologie, Hepatologie, Infektiologie und Ernährungsmedizin, Mannheim
  - Universitätsklinikum Marburg, Klinik für Innere Medizin, Gastroenterologie, Stoffwechsel und Endokrinologie, Marburg
  - Klinikum der Universität München, AG Onkologie der Med Klinik III, München
  - Klinikum Rechts der Isar der TU München, Klinik und Poliklinik für Chirurgie, München
  - Universitätsklinikum Regensburg, Klinik und Poliklinik für Chirurgie, Regensburg
  - Universitätsmedizin Rostock, Klinik III (Hämatologie, Onkologie, Palliativmedizin), Zentrum für Innere Medizin, Rostock
  - Caritasklinikum Saarbrücken St. Theresia, Saarbrücken
  - Universitätsklinikum Ulm, Klinik für Innere Medizin I Gastroenterologie-Endokrinologie-, Nephrologie-, Ernährung und Stoffwechselkrankheiten, Ulm
  - Universitätsklinikum Würzburg, Medizinische Klinik und Poliklinik II Zentrum für Innere Medizin, Würzburg
- Sweden (5):
  - Centralsjukhuset, Karlstad
  - Universitetssjukhuset, Linköping
  - Skånes universitetssjukhus, Lund
  - Norrlands universitetssjukhus, Umeå
  - Akademiska sjukhuset, Uppsala

IPD SHARING:
Plan to Share IPD: No